CLINICAL TRIAL: NCT01050699
Title: Sleep Intervention During Acute Lung Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sairam Parthasarathy, Associate Professor of Medicine, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC# 09-0232-01; 1R01HL095748-01A1 (NIH)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Critical Illness; Sleep; Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: critical illness; sleep; polysomnography; inflammatory cytokines; dexmedetomidine; acute lung injury; acute respiratory distress syndrome; midazolam; fentanyl; cytokines
MeSH Terms: conditions — Critical Illness; Acute Lung Injury; Respiratory Distress Syndrome | interventions — Dexmedetomidine; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine plus saline
  Interventions: Drug: Dexmedetomidine
- Usual Care (Active Comparator): Midazolam and Fentanyl
  Interventions: Drug: Midazolam and Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous continuous infusion will be initiated with a (optional) loading dose of 1 mcg/Kg over 10 minutes followed by a maintenance infusion of 0.5 mcg/kg/hour for 24 hours.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Midazolam and Fentanyl — Midazolam (Versed): Loading dose 2-4 mg IV bolus followed by continuous infusion at 1-7 mg/hour.
  Open label aliquots for pain (Midazolam 1- 4 mg IV bolus.)
  Fentanyl: Loading dose 50-200 mcg IV bolus; Continuous infusion rate 50-300 mcg/hour. Open label aliquots for pain (Fentanyl 50 - 200 mcg IV bolus.)
  Other Names: Versed (Midazolam); Fentanyl Citrate Injection, USP (Fentanyl)
  Arms: Usual Care

SUMMARY:
The central purpose of this proposal is to study the short-term effects of sedation with sympatholysis, using α2 adrenergic agent Dexmedetomidine, on sleep and inflammation in critically ill patients with Acute Lung Injury and Acute Respiratory Disorder Syndrome (ALI/ARDS). An additional objective is to determine the effect of Dexmedetomidine sedation on the in-vitro production of sleep-modulating inflammatory cytokines by peripheral blood mononuclear cells of critically ill patients with ALI/ARDS.

DETAILED DESCRIPTION:
Critically ill patients with acute lung injury and acute respiratory distress syndrome (ALI/ARDS) who receive mechanical ventilation can suffer from severe sleep disruption despite continuous sedative infusions. Sleep disruption, in turn, may activate the sympathetic nervous system and cause elevation of circulating inflammatory cytokines, which, in turn, may play a causative role in delirium and post-traumatic stress disorder through consolidation of unpleasant memories during awakenings from sleep. Currently, there is very little understanding of the inter-relationship between critical illness, sleep, and neuropsychological well-being, due to the lack of intervention-based trials that improve sleep during critical illness. The central purpose of this proposal is to study the short-term effects of sedation with sympatholysis (central α2 adrenergic agent) on sleep and inflammation in critically ill patients with ALI/ARDS. Sedation with sympatholysis will be achieved by a novel sleep-promoting agent with central α2 adrenergic properties. This FDA approved novel sedative agent, dexmedetomidine, has been shown to decrease delirium (an independent predictor of mortality) and decrease duration of mechanical ventilation and ICU stay in critically ill patients receiving mechanical ventilation (Riker et al, JAMA 2009;301:542-44 and Pandharipande et al, JAMA 2007;298:2644-53). We will undertake sleep studies and measure circulating inflammatory cytokines that modulate sleep in patients with ALI/ARDS randomized to receive two different sedation strategies: central α2 adrenergic sedative-analgesic (dexmedetomidine) versus a conventional sedation strategy (midazolam and fentanyl) in a randomized, double blind, cross-over study. Specific Aim 1: To assess the short-term effect of an α2 adrenergic agent on sleep quality in critically ill patients with ALI/ARDS. Specific Aim 2: To assess the short-term effect of an α2 adrenergic agent on sleep-modulating inflammatory cytokines in critically ill patients with ALI/ARDS. Specific aim 3: To determine the effect of α2 adrenergic agent on the in-vitro production of sleep-modulating inflammatory cytokines by peripheral blood mononuclear cells of patients with ALI/ARDS. Collectively, our study will identify whether sleep disruption in such patients can be minimized. In the long-term, this program of research will identify sedation practices that are least associated with adverse short- and long-term consequences of critical illness, and thereby ultimately help improve quality of life of patients surviving critical illness

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-85 (inclusive)
* Potential subjects receiving mechanical ventilation
* Potential subjects must have:

  1. Acute hypoxemia with a PaO2/FiO2 < 300 mm Hg (for ALI) OR < 200 mm Hg (for ARDS),
  2. Bilateral infiltrates (including very mild infiltrates)
  3. No clinical evidence of left atrial hypertension, or a pulmonary artery wedge pressure < 18 mm Hg.
* Potential subjects will be recruited after intubation and following a (systolic BP > 90 mm Hg on 2 or less continuous infusion of pressors) and ventilatory parameters (requiring < 60% fractional inspired O2 concentration [FiO2] and PEEP < 8 cm H2O).

Exclusion Criteria:

* Acute myocardial infarction or unstable angina or active myocardial ischemia
* Potential subjects who are considered too unstable to undergo this investigation by their primary physician.

  1. Symptomatic bradycardia (ventricular rate < 50 accompanied by hypotension [Systolic blood pressure < 90 mm Hg] or atrio-ventricular block [second degree type II or greater]).
  2. Known inability to tolerate beta-blockers or dexmedetomidine.
  3. Systolic blood pressure < 90 mmHg despite continuous infusions of 2 vasopressors before the start of study drug infusion.
* Potential subjects who are comatose or suffering from severe debilitating neurological disease (Intracerebral hemorrhage).
* History of severe dementia (derived from medical records or family sources).
* Active seizures
* Alcohol abuse by history
* Clinical evidence for decompensated congestive heart failure (elevated jugular venous distension, dependent edema) with echocardiographic evidence for significant systolic heart failure- left ventricular ejection fraction <30%.
* Renal failure (on renal dialysis); Hepatocellular failure (Child-Pugh class C).
* Metastatic or terminal cancer and patients with do-not-resuscitate orders
* Pregnancy
* Potential subjects who are expected to be extubated within 48 hours

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-08; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Specific Aim 1: To assess the short-term effect of an α2 adrenergic agent on sleep quality in critically ill patients with ALI/ARDS. | 72 hours

SECONDARY OUTCOMES:
Specific Aim 2: To assess the short-term effect of an α2 adrenergic agent on sleep-modulating inflammatory cytokines in critically ill patients with ALI/ARDS. | 72 hours
Specific aim 3: To determine the effect of α2 adrenergic agent on the in-vitro production of sleep-modulating inflammatory cytokines by peripheral blood mononuclear cells of patients with ALI/ARDS. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - University Medical Center, Tucson, Arizona